CLINICAL TRIAL: NCT03820362
Title: Personal Identity, Cognitive Factors and Psychotic Symptoms in Schizophrenia and Related Disorders: A Cross-sectional Study With the Repertory Grid Technique
Brief Title: The Role of Personal Identity in Psychotic Symptoms: a Study With the Repertory Grid Technique
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Agència de Gestió d'Ajuts Universitaris i de Recerca, Catalunya, Spain (Unknown); Ministerio de Educación y Formación Profesional, Spain (Unknown)
Responsible Party: Principal Investigator, Helena García Mieres, M.Sc., Ph.D. Cand., University of Barcelona
Other Study IDs: FPU15/01721
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia; Psychotic Disorders; Self
Keywords: personal identity; personal constructs
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Personal identity is being recently recognized as a core element for mental health disorders, with relevant clinical implications. However, scarcity of data exists on its role in schizophrenia and related disorders. The repertory grid (RGT), a technique derived from personal construct theory, has been used in different clinical and non-clinical contexts for the study of the construction perception of self and others, to appreciate aspects of interpersonal construing such as polarization and differentiation (unidimensional thinking) or self-construction.and Our study aims to explore the potential influence of the structure of personal identity and of other relevant cognitive factors (social cognition, metacognition, neurocognition) in positive and negative symptoms in people suffering schizophrenia and related disorders.

DETAILED DESCRIPTION:
Over recent years, the importance of the sense of self and personal identity in psychopathology and its treatment has been highlighted. Several studies inspired in the Personal Construct Psychology framework have found a variety of identity characteristics in clinical conditions such as depression or eating disorders, but the evidence in schizophrenia and other psychotic related disorders is scarce.

In addition, current psychological models of positive and negative symptoms highlight the influence of neurocognition, social cognition and self-concepts in the development and maintenance of psychotic experiences. Despite the recognized need of person-centered approaches to understand psychopathology processes in psychosis, psychological models for explaining psychotic symptoms have not explored sufficiently the role of this kind of person-centered measures.

Aim

1. To examine the influence of the structure of personal identity and other relevant cognitive factors in positive and negative symptoms

Hypotheses

1. Positive symptoms will be influenced by dichotomous thinking style and construction of self as measured with the RGT.
2. Negative symptoms will be affected by the richness of the construct system as measured with the RGT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia, psychotic disorder not otherwise specified, delusional disorder, schizoaffective disorder, brief psychotic disorder, or schizophreniform disorder
* age between 18 and 60 years.
* patients from outpatient mental health units

Exclusion Criteria:

* traumatic brain injury, dementia, or intellectual disability (pre-morbid IQ <70)
* current substance dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients recruited from the community, suffering schizophrenia and related disorder
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Self-ideal discrepancy, RGT | 2 hours
  Self-esteem. Possible range: 0-0,60. Higher values represent a worse outcome
Self-others discrepancy, RGT | 2 hours
  Perceived social isolation. Possible range: 0-0,60. Higher values represent a worse outcome
Interpersonal construct differentiation, RGT | 2 hours
  Percentage of Variance Accounted for the First Factor. Possible range: 0-100. Higher values represent a worse outcome
Polarization, RGT | 2 hours
  Dichotomous thinking style in the interpersonal context. Possible range: 0-100. Higher values represent a worse outcome
Number of elicited constructs, RGT | 2 hours
  Quantity of constructs that the person is able to express to describe self and others. Possible range: 10-50. Higher values represent a better outcome
Psychotic symptoms (PANSS, Kay et al. 1987; Peralta & Cuesta, 1994). | 40 minutes
  Positive and negative symptoms of psychosis. Range: 7-112. Higher values represent a worse outcome.
Metacognition: BCIS (Beck et al. 2004; Gutiérrez-Zotes et al. 2012); Garety et al, 1991; Dudley et al, 1997) | 15 minutes
  Cognitive insight. Range: 0-45. Higher values represent a better outcome
Theory of mind: the Hinting Task (Corcoran et al., 1995; Gil-Sanz et al., 2012) | 5 minutes
  Possible range: 0-12. Higher values represent a better outcome
General intellectual functioning (WAIS) | 20 minutes
  vocabulary subscale. Range: 70-140. Higher values represent a better outcome
Executive functioning: WSCT (Bergs et al., 1948) | 15 minutes
  Wisconsin Card Sorting Test. Categories completed and perseverative errors. Higher values represent a better outcome

SECONDARY OUTCOMES:
Sociodemographical data | 10 minutes
  Gender, chronicity, antipsychotic dosage, diagnosis, age, marital status, education level, employment situation
Depressive symptoms | 10 minutes
  Beck Depression Inventory (Beck et al. 1996; Sanz, Perdigón & Vázquez, 2003). Range_ 0-63. High values represent a worse outcome.
General functioning | 5 minutes
  Global Assessment of Functioning (Endicot et al., 1976). Range: 0-100. Higher values represent a better outcome.
Self-esteem | 5 minutes
  Rosenberg self-esteem scale (Martín Albó et al., 2007). Range: 0-40. Higher values represent a better outcome
Social functioning | 20 minutes
  Social Functioning Scale (Birchwood et al., 1990; Torres & Olivares, 2000). Range: Range: 45-195
Psychological distress | 10 minutes
  CORE-OM (Evans et al., 2002; Trujillo et al., 2016). Range: 0-4. Higher values represent a worse outcome
Jumping to Conclusions | 15 minutes
  The beads task (Garety et al., 1991; Dudley et al, 1997). Dichotomous: yes/no. A "yes" represents a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Helena García-Mieres, MsC, Principal Investigator — Universitat de Barcelona & Parc Sanitari Sant Joan de Déu; Susana Ochoa, PhD, Study Director — Parc Sanitari Sant Joan de Déu; Guillem Feixas, PhD, Study Director — University of Barcelona
Locations (1):
- Parc Sanitary Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided